CLINICAL TRIAL: NCT07120867
Title: Impact of Pleural Manometry on the Assessment and Treatment of Malignant Pleural Effusion: A Pilot Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-DPM-2022-133
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Malignant Pleural Effusions (Mpe)
MeSH Terms: conditions — Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Pleural Manometry) (No Intervention): Patients in this group will undergo standard management for malignant pleural effusion without pleural manometry. Therapeutic decisions such as pleurodesis or placement of a tunneled pleural catheter will be made based on clinical judgment and usual care protocols, without pleural pressure measurements.
- Pleural Manometry Group (Experimental): Patients in this group will undergo pleural manometry during the first thoracentesis. If pleural pressure measurements suggest that the lung expands, pleurodesis will be recommended. If the lung is non-expandable, pleurodesis will be avoided and a tunneled pleural catheter will be offered.
  Interventions: Diagnostic Test: Pleural manometry

INTERVENTIONS:
Diagnostic Test: Pleural manometry — Pleural manometry will be performed during the first thoracentesis using a water column connected to the pleural drainage system. Pleural pressure will be measured at baseline and at intervals during fluid removal to evaluate lung expandability. The water column manometer allows estimation of pressure changes in real time. Based on the pressure curve and indicators of non-expandable lung (such as early pressure drop, plateauing, or sustained negative pressures), the treatment plan will be adapted. If adequate lung re-expansion is observed, pleurodesis will be considered. If the pressure pattern suggests a non-expandable lung, pleurodesis will be avoided due to the high risk of failure, and a tunneled pleural catheter will be recommended instead.
  Arms: Pleural Manometry Group

SUMMARY:
The goal of this clinical trial is to find out if performing a pleural fluid drainage (thoracentesis) together with the measurement of pressure inside the chest (pleural manometry) during the same procedure can help doctors choose the best treatment for each patient with malignant pleural effusion.The main questions it aims to answer are:

* Is the use of pleural manometry associated with a higher success rate in managing malignant pleural effusion through pleurodesis?
* Can the use of pleural manometry help guide optimal therapeutic decision-making in malignant pleural effusion?

Researchers will compare the success of the chosen treatment in patients who undergo pleural manometry to those who do not, to see if pleural manometry helps improve treatment outcomes for malignant pleural effusion.

Participants will:

* Receive treatment according to the hospital's standard clinical practice for managing malignant pleural effusion.
* If assigned to the manometry group, they will undergo pleural manometry during their first thoracentesis.
* If the manometry results suggest that the lung can fully expand, they will be referred for pleurodesis-just as patients in the non-manometry group are.
* If the manometry results suggest that the lung cannot fully expand, pleurodesis will not be recommended due to the high risk of failure. Instead, placement of a tunneled pleural catheter will be advised to help control symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer and symptomatic patient with at least one of the following:

  * Malignant pleural effusion confirmed by cytology.
  * Recurrent exudative pleural effusion without an alternative diagnosis in the context of confirmed extrapleural cancer.
  * Pleural effusion associated with hypermetabolic pleural thickening suggestive of malignant pleural effusion.

Exclusion Criteria:

* Radiological evidence of non-expandable lung
* Life expectancy <1 month (LENT score: high risk)
* Previous ipsilateral lobectomy or pneumonectomy
* Previous ipsilateral chemotherapy or radiotherapy
* Presence of infected pleural effusion
* Patient preference for tunneled pleural catheter placement
* Pregnancy
* Thrombocytopenia or coagulopathy
* Contraindication to general anesthesia or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Successful pleurodesis based on radiographic assessment | 30 days after hospital discharge
  Number of participants with successful pleurodesis, defined as absence of recurrent pleural effusion or presence of minimal or loculated effusion that does not require additional therapeutic procedures to relieve symptoms. Assessment will be performed using chest X-ray interpreted by the thoracic surgeon at the follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreiro L, San Jose E, Gude F, Valdes L. Pleural Fluid Analysis and Pleural Elastance as Predictors of Response to Pleurodesis in Patients With Malignant Pleural Effusion. Arch Bronconeumol (Engl Ed). 2018 Mar;54(3):163-165. doi: 10.1016/j.arbres.2017.07.020. Epub 2017 Sep 18. No abstract available. English, Spanish. PMID 28927859
- [Background] Lan RS, Lo SK, Chuang ML, Yang CT, Tsao TC, Lee CH. Elastance of the pleural space: a predictor for the outcome of pleurodesis in patients with malignant pleural effusion. Ann Intern Med. 1997 May 15;126(10):768-74. doi: 10.7326/0003-4819-126-10-199705150-00003. PMID 9148649
- [Background] Huggins JT, Doelken P. Pleural manometry. Clin Chest Med. 2006 Jun;27(2):229-40. doi: 10.1016/j.ccm.2005.12.007. PMID 16716815
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691